CLINICAL TRIAL: NCT06313736
Title: How Long Should a Behavioral Activation Single-session Intervention be? A Four-armed Trial Comparing Effectiveness by Intervention Duration
Brief Title: What SSI Duration is Most Effective? An Online Experiment With American Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jessica Schleider, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00220591_shortening; 2T32MH115882-06A1 (NIH)
Record Dates: First submitted 2024-03-11; First posted 2024-03-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Depression
Keywords: Single-session intervention; Length; Duration; Effectiveness; Active elements
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of four different conditions.
Who Masked: Participant, Investigator
Masking Description: Participants will be aware that they will be assigned to an intervention designed to help them with depressive symptoms. They will know that the study compares multiple interventions but will not know to which arm they have been assigned. Additionally, the measures will be self-administered, so there is no scope for evaluator bias. There will be no interaction between participants and investigators.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 15-minute single-session depression intervention (Experimental): This is the adult version of the Action Brings Change (ABC) Project.
  Interventions: Behavioral: Action Brings Change Project (15-minute adult version)
- 10-minute single-session depression intervention (Experimental): This includes a shortened version of the ABC Project.
  Interventions: Behavioral: Action Brings Change Project (10-minute adult version)
- 6-minute single-session depression intervention (Experimental): This includes a shortened version of the ABC Project.
  Interventions: Behavioral: Action Brings Change Project (6-minute adult version)
- 2-minute single-session depression intervention (Experimental): This includes a shortened version of the ABC Project.
  Interventions: Behavioral: Action Brings Change Project (2-minute adult version)

INTERVENTIONS:
Behavioral: Action Brings Change Project (15-minute adult version) — The ABC Project is a self-guided online single-session intervention based on principles of behavioral activation. In a slightly different form intended for adolescents, it has demonstrated efficacy in several studies. Its adult version has also shown some efficacy.
  Other Names: ABC Project (15-min)
  Arms: 15-minute single-session depression intervention
Behavioral: Action Brings Change Project (10-minute adult version) — This is a 10-minute shortened version of the 15-minute adult version of the ABC Project. The research team created it and pilot-tested it.
  Other Names: ABC Project (10-min)
  Arms: 10-minute single-session depression intervention
Behavioral: Action Brings Change Project (6-minute adult version) — This is a 6-minute shortened version of the 15-minute adult version of the ABC Project. The research team created it and pilot-tested it.
  Other Names: ABC Project (6-min)
  Arms: 6-minute single-session depression intervention
Behavioral: Action Brings Change Project (2-minute adult version) — This is a 2-minute shortened version of the 15-minute adult version of the ABC Project. The research team created it and pilot-tested it.
  Other Names: ABC Project (2-min)
  Arms: 2-minute single-session depression intervention

SUMMARY:
In a previous study (https://osf.io/qdznc), the research team found that an 8-minute version of a single-session intervention for loneliness was more effective than a 23-minute version of it. The present work aims to further explore the relationship between intervention duration and effectiveness.

In this online trial, participants will be randomized to a 15-minute single-session depression intervention called the Action Brings Change (ABC) Program, a 10-minute version of it, a 6-minute version of it, or a 2-minute version of it. The main analysis will evaluate how change in depressive symptoms over eight weeks differs across conditions.

ELIGIBILITY:
Inclusion Criteria: Participants must be:

* Located in the United States
* At least 18 years old
* Patient Health Questionnaire-8 (PHQ-8) score of at least 10 (moderate or more severe) at screener.
* Able to read and speak fluent English
* Able to access to the internet via a computer, tablet or smartphone for the next eight weeks

Exclusion Criteria:

* Participants who have completed the first session of the study before or completed another study testing a depression intervention from our laboratory via the same participant recruitment platform in the past two months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1145 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-8 at 8 weeks (PHQ-8; Kroenke et al., 2009) | Baseline to 8 weeks post-intervention
  Patient Health Questionnaire-8 is a well-validated and self-administered measure to assess depression symptom severity in the general population. Participants are asked to rate how often they are bothered by 8 items (e.g., Poor appetite or overeating) on a scale of 0 (Not at all) to 3 (Nearly every day). Total score can range from 0 to 24, with higher scores indicating higher symptom severity.

SECONDARY OUTCOMES:
Change in Beck Hopelessness Scale at 8 weeks (BHS-4; Perczel Forintos et al., 2013) | Baseline to 8 weeks post-intervention
  Beck Hopelessness Scale-4 is the 4-item version of the 20-item Beck Hopelessness scale (Beck et al. 1974). Participants will be asked to rate 4 items assessing different aspects of hopelessness (e.g., My future seems dark to me) on a scale of 0 (Absolutely disagree) to 3 (Absolutely agree). Total score can range between 0 to 12 with higher scores indicating higher hopelessness.
Change in Beck Hopelessness Scale - 4-item at post-intervention | Baseline to immediately post-intervention
  Beck Hopelessness Scale-4 is the 4-item version of the 20-item Beck Hopelessness scale (Beck et al. 1974). Participants will be asked to rate 4 items assessing different aspects of hopelessness (e.g., My future seems dark to me) on a scale of 0 (Absolutely disagree) to 3 (Absolutely agree). Total score can range between 0 to 12 with higher scores indicating higher hopelessness.
Change in UCLA Loneliness Scale 3-item version at 8-week follow-up (ULS-3; Hughes et al., 2004) | Baseline to 8 weeks post-intervention
  The ULS-3 is the 3-item version of the 20-item UCLA Loneliness Scale. The measure includes questions such as "how often do you feel left out" with responses ranging from 1 (hardly ever) to 3 (often), producing a total score between 3 and 9. Researchers have labeled people who score 3-5 as "not lonely" and those who score 6-9 as "lonely."
Presence of an "Aha! moment" at post-intervention | Immediately post-intervention
  The survey will ask participants if they experienced an "Aha! moment" during the SSI.
Presence of an "Aha! moment" at 8 weeks post-intervention | 8 weeks post-intervention
  The survey will ask participants if they experienced an "Aha! moment" during the SSI.
Significance of the "Aha! moment" at immediately post-intervention | Immediately post-intervention
  Among participants who report an Aha! Moment, the survey will ask how significant they felt that Aha! was (on a scale from 1 [not at all significant] - 5 [extremely significant]).
Significance of the "Aha! moment" at 8 weeks post-intervention | 8 weeks post-intervention
  Among participants who report an Aha! Moment, the survey will ask how significant they felt that Aha! was (on a scale from 1 [not at all significant] - 5 [extremely significant]).
Change in Frequency of actions and thoughts scale at post-test at 8 weeks post-intervention (FATS; Terides et al., 2016) | Baseline to 8 weeks post-intervention
  A 12-item measure of adaptive thoughts and behaviors, improvement in which might be a target of cognitive behavioral therapy. Range 0-48 with higher scores indicating greater frequency of adaptive thoughts and behaviors.
Expected improvement at post-intervention (from the Credibility / Expectancy Questionnaire; Devilly, 2004) | Immediately post-intervention
  This will be computed as the sum of two items: "At this point, how successful do you think this treatment will be in reducing your feelings of depression?" and "Over the next few weeks, how much improvement in your feelings of depression do you think will occur?"). Each item will be rated from 1-9 and will be summed together to create a total score of 2-18 with higher scores indicating greater expected improvement.
Self-reported improvement at 8-weeks post-intervention (adapted from the Credibility/ Expectancy Questionnaire; Devilly, 2004) | 8 weeks post-intervention
  This will be computed as the sum of two items: "At this point, how successful do you think this treatment was in reducing your feelings of depression?" and "Over the past eight weeks, how much improvement in your feelings of depression do you think occurred?"). Each item will be rated from 1-9 and will be summed together to create a total score of 2-18 with higher scores indicating greater improvement.
Intervention satisfaction star rating at post-intervention | Immediately post-intervention
  The survey will evaluate participants' satisfaction with the intervention they completed using a star rating from 1 to 5 stars, with 1 star indicating very low satisfaction and 5 stars indicating very high satisfaction.
Intervention satisfaction star rating at 8 week follow-up | 8 weeks post-intervention
  The survey will evaluate participants' satisfaction with the intervention they completed using a star rating from 1 to 5 stars, with 1 star indicating very low satisfaction and 5 stars indicating very high satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica L Schleider, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Medical Social Sciences, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available once they are anonymized and all the planned analyses have been completed by the investigators.
Supporting Information: SAP, Analytic Code
Time Frame: Anonymized data and code will be made publicly available here (https://osf.io/g846j/) upon publication of trial results.
Access Criteria: Publicly available

REFERENCES:
- [Background] Schleider JL, Mullarkey MC, Fox KR, Dobias ML, Shroff A, Hart EA, Roulston CA. A randomized trial of online single-session interventions for adolescent depression during COVID-19. Nat Hum Behav. 2022 Feb;6(2):258-268. doi: 10.1038/s41562-021-01235-0. Epub 2021 Dec 9. PMID 34887544
- [Background] Kroenke K, Strine TW, Spitzer RL, Williams JB, Berry JT, Mokdad AH. The PHQ-8 as a measure of current depression in the general population. J Affect Disord. 2009 Apr;114(1-3):163-73. doi: 10.1016/j.jad.2008.06.026. Epub 2008 Aug 27. PMID 18752852
- [Background] Perczel Forintos D, Rozsa S, Pilling J, Kopp M. Proposal for a short version of the Beck Hopelessness Scale based on a national representative survey in Hungary. Community Ment Health J. 2013 Dec;49(6):822-30. doi: 10.1007/s10597-013-9619-1. Epub 2013 Jun 12. PMID 23756722
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Terides MD, Dear BF, Karin E, Jones MP, Gandy M, Fogliati VJ, Kayrouz R, Staples LG, Titov N. The frequency of actions and thoughts scale: development and psychometric validation of a measure of adaptive behaviours and cognitions. Cogn Behav Ther. 2016 Apr;45(3):196-216. doi: 10.1080/16506073.2016.1149876. Epub 2016 Feb 29. PMID 26926484
- [Background] Hughes ME, Waite LJ, Hawkley LC, Cacioppo JT. A Short Scale for Measuring Loneliness in Large Surveys: Results From Two Population-Based Studies. Res Aging. 2004;26(6):655-672. doi: 10.1177/0164027504268574. PMID 18504506

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-17): https://cdn.clinicaltrials.gov/large-docs/36/NCT06313736/Prot_SAP_000.pdf